CLINICAL TRIAL: NCT04256681
Title: SNAP: Measurement of the Subjective Perception of the Symptom in Hereditary Spastic Paraparesis (HSP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Eugenio Medea (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: GIP 595
Record Dates: First submitted 2020-02-03; First posted 2020-02-05 (Actual); Last update posted 2021-11-26 (Actual); Status verified 2021-11

CONDITIONS: Hereditary Spastic Paraparesis
Keywords: OUTCOME MEASURE, HEREDITARY SPASTIC PARAPLEGIA
MeSH Terms: conditions — Spastic Paraplegia, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients affected by hereditary spastic paraplegia (Experimental): 40 subjects affected by genetically determined hereditary spastic paraparesis or subjects without defined genetics but who unequivocally show a dominant or recessive familiarity with exclusive involvement of the pyramidal system.
  Interventions: Other: SNAP questionnaire
- healthy subjects (Active Comparator): 40 healthy subjects will also be recruited to whom the questionnaire will be submitted to assess the variability of the score within a healthy population.
  Interventions: Other: SNAP questionnaire

INTERVENTIONS:
Other: SNAP questionnaire — The SNAP questionnaire will be administered 2 times in 2 consecutive days to evaluate its reliability. The questionnaire will be self-filled by the patient. Then the SPRS scale and, where possible, the 6MWT will be administered.

SUMMARY:
The Self-Notion and Perception (SNAP) questionnaire developed at IRCCS E.Medea by Eleonora Diella and Roberta Morganti, arises from the need to quantify the subjective perception of the patient suffering from HSP of the typical symptoms of pathology, such as spasticity, weakness, changes in balance, resistance in walking, pain and fatigue. The purpose of this study is to validate this instrument and test its reliability, looking for correlations with the measurement scales used in the literature for the evaluation of the patient with HSP. The most used for this population are the Spastic Paraplegia Rating Scale (SPRS) and the Six-Minute Walk Test (6MWT) which assess the severity of the disease and the level of endurance (8-9) respectively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of genetically determined hereditary spastic paraparesis or subjects without defined genetics but who unequivocally show at the time of evaluation a dominant or recessive familiarity with exclusive involvement of the pyramidal system
* age> 9 years
* IQ> 80
* The patient must be able to walk for at least 10 meters. Indoors, even with help

Exclusion Criteria:

* Age less than 9 years
* IQ <80,
* loss of gait
* psychopathological aspects that can affect the validity of the data collected

Min Age: 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2018-10-30 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Test the validity, investigating the correlation with Spastic Paraplegia Rating Scale and with Six-Minute Walk Test, and the reliability (through test-retest mode) of the SNAP questionnaire in the aforementioned population. | 2 days
  the Spastic Paraplegia Rating Scale (SPRS) and the Six-Minute Walk Test (6MWT) which assess the severity of the disease and the level of endurance respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Eleonora Diella, Bosisio Parini, Italy

REFERENCES:
- [Derived] Diella E, D'Angelo MG, Stefan C, Girardi G, Morganti R, Martinuzzi A, Biffi E. Validation of the Italian version of a patient-reported outcome measure for Hereditary Spastic Paraplegia. PLoS One. 2024 Apr 1;19(4):e0301452. doi: 10.1371/journal.pone.0301452. eCollection 2024. PMID 38557877